CLINICAL TRIAL: NCT00785395
Title: Up-down Determination of the ED90 of Oxytocin Infusions for the Prevention of Postpartum Uterine Atony in Parturients Undergoing Cesarean Delivery
Brief Title: Up-Down Oxytocin Infusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Ronald George, Primary Investigator, MD, FRCPC, Assistant Professor, IWK Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IWK-4329-2008
Record Dates: First submitted 2008-10-27; First posted 2008-11-05 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2008-11

CONDITIONS: Uterine Atony
MeSH Terms: conditions — Uterine Inertia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Oxytocin infusion

INTERVENTIONS:
Drug: Oxytocin infusion — Up-down dosing determination

SUMMARY:
This study is designed to determine the minimum effective dose (ED90) of infusions of oxytocin for the prevention of uterine atony / postpartum hemorrhage and the need for additional uterotonics, in low risk parturients presenting for an elective CD.

The primary outcome measure is the response of effective uterine contraction as either satisfactory or unsatisfactory as determined by the obstetrician blinded to the oxytocin infusion dose. Secondary outcomes will include need for additional uterotonics, calculated intra-operative blood loss and presence of oxytocin related adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Non-emergent cesarean delivery with planned spinal anesthesia (i.e. elective planned cesarean delivery for malposition, patient choice, cervical pelvic disproportion, previous cesarean delivery and other diagnosis that require a predetermined cesarean delivery)
2. American Society of Anesthesia physical status class I & II (ASA I - Healthy, ASA II - mild and controlled systemic disease, eg. controlled essential hypertension)
3. Age ≥ 18 years
4. Term gestational age (≥ 37 weeks)
5. English-speaking

Exclusion Criteria:

1. Morbid Obesity (Body Mass Index ≥ 45 kg/m2) (Morbidly obese parturients require a dose of local anesthetic less than the standardized dose in this study and the blood pressure cuff occasionally needs to be replaced by an intraarterial catheter due to limitations in size)
2. Laboring women
3. Urgent or emergency cesarean delivery
4. Severe hypertensive disease of pregnancy defined as systolic blood pressure (SBP) > 160mmHg, diastolic blood pressure (DBP) > 110mmHg and/or requiring antihypertensive treatment or associated with significant proteinuria
5. Severe maternal cardiac disease
6. Subjects predisposed to uterine atony and postpartum hemorrhage (i.e. placenta previa, multiple gestation, macrosomia, polyhydramnios, uterine abnormalities, or bleeding diathesis, > 2 previous CD)
7. Fetal anomalies /Intrauterine Fetal Demise
8. Failed spinal anesthesia
9. Patient enrollment in another study involving a study medication within 30 days of CD
10. Any other physical or psychiatric condition which may impair their ability to cooperate with study data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the response of effective uterine contraction as either satisfactory or unsatisfactory as determined by the obstetrician blinded to the oxytocin infusion dose. | 3 minutes

SECONDARY OUTCOMES:
Secondary outcomes will include need for additional uterotonics, calculated intra-operative blood loss and presence of oxytocin related adverse effects. | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B George, MD FRCPC, Principal Investigator — IWK
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] George RB, McKeen D, Chaplin AC, McLeod L. Up-down determination of the ED(90) of oxytocin infusions for the prevention of postpartum uterine atony in parturients undergoing Cesarean delivery. Can J Anaesth. 2010 Jun;57(6):578-82. doi: 10.1007/s12630-010-9297-1. Epub 2010 Mar 18. PMID 20238255